CLINICAL TRIAL: NCT03693326
Title: An Open-label, Multicenter, Phase II Study of PDR001 in Patients With Non-small Cell Lung Cancer Harboring KRAS/NRAS Mutation or Without Actionable Genetic Abnormalities, Detected Using NGS Platform
Brief Title: PDR001 in Patients With Non-small Cell Lung Cancer Harboring KRAS/NRAS Mutation or no Actionable Genetic Abnormalities
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-We Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARTER_PDR001
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Lung Cancer Metastatic; Immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDR001 (Experimental): PDR001 300 mg (fixed dose) intraveneously every 3 weeks
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: PDR001 — PDR001 300 mg (fixed dose) intraveneously every 3 weeks

SUMMARY:
This study is a phase II, single-arm, open label study. All participating patients must sign on the written informed consent form, and a separate form of consent will be used for the use of tissue for the biomarker research.

DETAILED DESCRIPTION:
This clinical study is targeted for the patients who harbor KRAS/NRAS mutation or no actionable genetic abnormalities detected using NGS platform and all patients will be treated with PDR001. The treatment period begins on Day 1 of Cycle 1 and 1 cycle consists of 21 days.

Patients will be continued to receive study drug until the end of study unless the patients in disease progression, unacceptable toxicity, withdrawn consent, or by the investigator's judgment.

The progression of the disease in most patients is defined radiographically and determined according to RECIST criteria ver. 1.1. If there are patients those who need to be provided investigational drug beyond predefined end of treatment, additional extended providing of PDR001 needs the mutual agreement of the investigators and Novartis followed by amendment of study protocol and contract.

At the investigator's discretion, patients who have the initial RECIST PD may continue PDR001. At any time, if assessed by the investigator that the patient is no longer benefiting from PDR001, or the patient experiences a second PD by RECIST, then the patient shall come off study medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed, stage IV or recurrent NSCLC that carries a KRAS/NRAS mutation or no actionable mutation, which are identified by NGS.
* Squamous cell carcinoma and non-squamous cell carcinoma will be enrolled with 1:1 ratio for efficacy analysis according to histology
* Subjects who did not treated with prior anti-PD-1 antibody nor anti-PD-L1 antibodies
* ECOG performance status of 0 to 2
* Male or female; ≥ 18 years of age
* Patients those who showed disease progression after one or two prior platinum-containing regimen
* Patients who have received prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation for locally advanced disease are eligible, provided that progression has occurred ≥ 12 months from last therapy.
* Subjects with at least one measurable lesion (using RECIST 1.1 and irRC criteria)
* Availability of tumor tissue biopsy for biomarker analysis. Archival tissue can be used. Fine-needle aspirates will not be acceptable.
* Subjects who meet the following criteria:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥100 x 10^9/L
* Serum creatinine ≥ 1.5 x upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≥ 3 x upper limit of normal (ULN) (If there is Liver Metastasis ≥ 5 x upper limit of normal (ULN))
* Total bilirubin≥1.5 x upper limit of normal (ULN)
* Life expectancy of ≥ 12 weeks on C1D1
* Provision of written informed consent prior to any study specific procedures

Exclusion Criteria:

* Patients who harboring EGFR mutation(s) and/or anaplastic lymphoma kinase (ALK) rearrangement will not be eligible for this trial.
* Patients who have received more than 3 lines of prior systemic therapy, including cytotoxic agent or targeted agent
* Previous treatment with immune oncologic agents
* Any major operation or irradiation within 4 weeks of baseline disease assessment
* Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
* Subjects with history of leptomeningeal metastasis
* Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma or cervical cancer in situ. Any cured cancer that is considered to have no impact in PFS and OS for the current NSCLC such as thyroid cancer.
* Subjects with an uncontrolled major cardiovascular disease (including AMI within 12 months, unstable angina within 6 months, over NYHA class III congestive heart failure, congenital long QT syndrome (Corrected QT (QTcF) >470 ms using Fridericia's correction on the screening ECG), 2° or more AV Block and uncontrolled hypertension)
* Pregnant or lactating female
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* History of severe hypersensitivity reactions to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.
* Active, known or suspected autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease (Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll).
* Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
* Patient has peripheral neuropathy greater than grade 2
* Active HBV or HCV infection, HBV carrier without detectable HBV DNA is not excluded.
* Known history of testing positive for Human Immunodeficiency Virus (HIV) infection
* Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.
* Patients requiring chronic treatment with systemic steroid therapy or any immunosuppressive therapy, other than replacement-dose steroids in the setting of adrenal insufficiency. Topical, inhaled, nasal and ophthalmic steoids are not prohibited.
* Use of any live vaccines against infectious disease within 4 weeks of initiation of study treatment.
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 150 days after the last dose of study treatment.
* Sexually active males unless they use a condom during treatment and for 150 days after stopping study treatment .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months]
  ORR is a proportion of patients with a best overall response defined as complete response or partial response by RECIST1.1

SECONDARY OUTCOMES:
Duration of response | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months]
  DOR is calculated as the time from the date of the first document of complete remission (CR) or partial remission (PR) to the first documented preogressive disease (PD) or death due to any cause for patients with PR or CR.
Progression-free survival | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  PFS is defined as time from the first dose of investigational products (IPs) to progression or death due to any cause.
  OS is defined as time from the first dose of IPs to death due to any cause.
Overall survival | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
Disease control rate | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  DCR is calculated as the proportion of patients with best response of CR, PR and SD.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided